CLINICAL TRIAL: NCT01746095
Title: A Phase 2, Randomized, Double Blind, Placebo-controlled Study of AeroVanc for the Treatment of Persistent Methicillin-resistant Staphylococcus Aureus Lung Infection in Cystic Fibrosis Patients
Brief Title: Efficacy and Safety Study of AeroVanc for the Treatment of Persistent MRSA Lung Infection in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Collaborators: Synteract, Inc. (Industry); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAV005-02
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; MRSA; Methicillin-resistant Staphylococcus aureus; Lung infection; AeroVanc; Vancomycin
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomycin hydrochloride inhalation powder (Experimental): 32 or 64 mg twice daily (BID)
  Interventions: Drug: Vancomycin hydrochloride inhalation powder
- Placebo inhalation powder (Placebo Comparator): Matching placebo inhalation powder BID
  Interventions: Drug: Placebo inhalation powder

INTERVENTIONS:
Drug: Vancomycin hydrochloride inhalation powder — There will be two treatment cohorts in this study, each comprised of 40 randomized (1:1 active to placebo) and treated patients (adults ≥18 and children ≥12 years of age). In Cohort 1, patients will be enrolled and randomized to receive the 32 mg dose of AeroVanc bid or placebo bid. Prior to starting enrollment in Cohort 2, a safety evaluation will be carried out by the Data Monitoring Committee (DMC) based on treatment data from the first 20 patients in Cohort 1. Subject to the Sponsor's written communication of the DMC's opinion of acceptable safety, the dose for the active arm in Cohort 2 will be escalated to 64 mg bid. Optionally, the active arm for Cohort 2 may also be kept the same (32 mg bid), or reduced to 16 mg bid, depending on the outcome of the DMC's safety evaluation.
  Other Names: AeroVanc
  Arms: Vancomycin hydrochloride inhalation powder
Drug: Placebo inhalation powder
  Arms: Placebo inhalation powder

SUMMARY:
The purpose of this study is to determine whether AeroVanc treatment is safe and effective in reducing the number of MRSA colony forming units in the lungs of cystic fibrosis patients.

DETAILED DESCRIPTION:
This is a Phase 2a randomized, multicenter, double-blind, placebo-controlled, parallel group study to examine the safety and efficacy of AeroVanc in the treatment of persistent MRSA lung infection in CF patients. Pharmacokinetics will be evaluated in a subgroup by measuring plasma and sputum concentrations of vancomycin.

Prior to treatment, patients will be randomized to receive either AeroVanc twice daily (bid), or placebo bid. Patients will be stratified based on the presence of a Pseudomonas aeruginosa (P. aeruginosa) co-infection that is being treated with a chronic suppression regimen. Patients with P. aeruginosa co-infection can be on any chronic inhaled suppression regimen (or nothing if the patient is considered stable in the opinion of the investigator despite the lack of treatment). Regardless of treatment regimen, if there is an off month, screening should be scheduled so that AeroVanc or placebo administration can be given during this time. Patients with no off month should be screened so that the AeroVanc or placebo administration period coincides with a treatment cycle other than TOBI (e.g., Cayston or colistin). All patients must have at least a 24-hour washout period after stopping their anti-Pseudomonas therapy and prior to the Visit 2 (Baseline) pre-dose microbiology sputum sample. The AeroVanc or placebo treatment duration is 28 days, during which efficacy and safety parameters will be measured, and after which patients will be followed up for 56 days.

There will be two treatment cohorts in this study, each comprised of 40 randomized (1:1 active to placebo) and treated patients (adults ≥18 and children ≥12 years of age). In Cohort 1, patients will be enrolled and randomized to receive the 32 mg dose of AeroVanc bid or placebo bid. Prior to starting enrollment in Cohort 2, a safety evaluation will be carried out by the Data Monitoring Committee (DMC) based on treatment data from the first 20 patients in Cohort 1. Subject to the Sponsor's written communication of the DMC's opinion of acceptable safety, the dose for the active arm in Cohort 2 will be escalated to 64 mg bid. Optionally, the active arm for Cohort 2 may also be kept the same (32 mg bid), or reduced to 16 mg bid, depending on the outcome of the DMC's safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old (and the legally authorized representatives of children ≥12 but <18 years old): Able to communicate with site personnel and to understand and voluntarily sign the Informed Consent Form (ICF). Children ≥12 but <18 years old: Able to communicate with site personnel and to understand and voluntarily sign the Assent Form.
2. Able and willing to comply with the protocol, including availability for all scheduled study visits.
3. Have a confirmed diagnosis of CF, determined by having clinical features consistent with the CF phenotype, plus one of the following: a) Positive sweat chloride test (value ≥60 mEq/L), or b) Genotype with two mutations consistent with CF (ie, a mutation in each of the cystic fibrosis transmembrane conductance regulator [CFTR] genes).
4. Be ≥12 years old at time of ICF/Assent Form signing.
5. Have sputum culture positive for MRSA at Screening, with at least 10,000 CFUs/mL of MRSA.
6. In addition to the screening sample, have at least two historical respiratory tract cultures (i.e., sputum and/or throat swab) positive for MRSA prior to Screening and evidence that the MRSA lung infection has persisted for at least 6 months prior to Screening.
7. Have forced expiratory volume in 1 second (FEV1) ≥30% and ≤100% of predicted that is normalized for age, gender, and height at Screening.
8. Evidence, defined as one or both of the following, that the persistent MRSA lung infection is suspected to be causing health consequences.

   * Have had at least one episode of acute pulmonary infection treated with non-maintenance antibiotics within 12 months from Screening. Initiation of treatment with intermittent inhaled anti-Pseudomonas therapy will not qualify as treatment with non-maintenance antibiotics.
   * Requires anti-MRSA treatment as part of a maintenance regimen to prevent pulmonary exacerbations or other respiratory symptoms.
9. Be able to perform all the techniques necessary to use the AeroVanc inhaler and measure lung function.
10. Be able to produce expectorated sputum samples or be able and willing to undergo standardized sputum induction.
11. Agree not to smoke from Screening through the end of the study.
12. Female patients of child-bearing potential are eligible to participate in this study only if they are NOT pregnant or lactating, and if the patient is using a highly effective method of birth control.
13. Patients with P. aeruginosa co-infection must either be stable on a regular suppression regimen of inhaled antibiotics or must be, in the opinion of the investigator, stable despite the lack of such treatment. Patients on a Cayston based therapy must have received at least 2 cycles of Cayston prior to Baseline (can be 2 consecutive months or 2 cycles over 4 months).

Exclusion Criteria:

1. Administration of any investigational drug or device within 28 days prior to ICF/Assent Form signing.
2. Use of iv or inhaled anti-MRSA drugs within 28 days or oral anti-MRSA drugs within 14 days prior to Visit 2 (ie, randomization, Baseline and AeroVanc/placebo treatment initiation).
3. A history of previous allergies or sensitivity to vancomycin, or other component(s) of the study drug or placebo except for a history of red-man syndrome.
4. History of severe cough/bronchospasm upon inhalation of dry powder inhalation product, or nebulized vancomycin.
5. Resistance to vancomycin at Screening (vancomycin resistant Staphylococcus aureus [VRSA], or vancomycin intermediate resistant Staphylococcus aureus [VISA], with minimum inhibitory concentration [MIC] ≥4 mcg/mL).
6. Oral corticosteroids in doses exceeding 10 mg prednisone per day or 20 mg prednisone every other day, or equipotent doses of another corticosteroid.
7. History of sputum culture or throat swab culture yielding B. cepacia or gladioli in the previous two years, or nontuberculosis mycobacteria in the previous six months.
8. An acute upper or lower respiratory infection, or pulmonary exacerbation within 7 days prior to Randomization.
9. Changes in antimicrobial, bronchodilator, anti-inflammatory or corticosteroid medications within 7 days prior to ICF/Assent Form signing.
10. Current daily continuous oxygen supplementation or requirement for more than 2 L/min at night.
11. Changes in physiotherapy technique or schedule within 7 days prior to ICF/Assent Form signing.
12. History of lung or other solid organ transplantation or currently on the list to receive lung or other solid organ transplantation.
13. A chest X-Ray at Screening with abnormalities indicating a significant acute finding (eg, pneumothorax, or pleural effusion).
14. Lactating female or female with a positive pregnancy test result. All women of childbearing potential will be tested.
15. Renal insufficiency, defined as creatinine clearance <50 mL/min using the Cockcroft-Gault equation for adults or Schwartz equation in children, at Screening.
16. Diagnosed with clinically significant hearing loss.
17. Abnormal liver function, defined as ≥4x upper limit of normal (ULN), of serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT), or known cirrhosis at the time of Screening.
18. Serum hematology or chemistry screening results which in the judgment of the Investigator would interfere with completion of the study.
19. Positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
20. Other findings or medical history at screening that, in the Investigator's opinion, would compromise the safety of the patient or the quality of the study data.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Dasenbrook, M.D., MHS, Principal Investigator — Case Western Reserve University School of Medicine and Rainbow Babies and Children's Hospital
Locations (38):
- United States (38):
  - Pulmonary Associates of Mobile, Mobile, Alabama
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Division of Pediatric Pulmonology, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Nemours Children's Clinic and Hospital, Orlando, Florida
  - New Lung Associates, PA; Lung Transplant, Adult Cystic Fibrosis, and the Center for Advanced Lung Diseases, Tampa General Hospital, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Cystic Fibrosis Clinic, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital Pediatric Cystic Fibrosis Center, Boston, Massachusetts
  - Boston Children's Hospital Cystic Fibrosis Center, Boston, Massachusetts
  - Wayne State University, Harper Hospital, Children's Hospital of Michigan, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Hofstra North Shore - Long Island Jewish School of Medicine, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rainbow Babies and Children's Hospital / University Hospitals Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine and Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Intermountain Cystic Fibrosis Center, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Lo DK, Muhlebach MS, Smyth AR. Interventions for the eradication of meticillin-resistant Staphylococcus aureus (MRSA) in people with cystic fibrosis. Cochrane Database Syst Rev. 2022 Dec 13;12(12):CD009650. doi: 10.1002/14651858.CD009650.pub5. PMID 36511181

RESULTS

PARTICIPANT FLOW:
Groups:
- AeroVanc 32 mg: Vancomycin hydrochloride inhalation powder 32 mg BID
- Placebo to 32 mg; Placebo to 64 mg: Placebo inhalation powder BID
- AeroVanc 64 mg: Vancomycin hydrochloride inhalation powder 64 mg BID
Period: Overall Study
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Started | 20 | 20 | 24 | 23
Completed | 16 | 16 | 11 | 15
Not Completed | 4 | 4 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg | Total
Number analyzed (Participants) | 20 | 20 | 24 | 23 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 4 | 4 | 21
  Between 18 and 65 years | 13 | 14 | 20 | 19 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 9 | 8 | 39
  Male | 7 | 11 | 15 | 15 | 48
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 24 | 23 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MRSA Sputum Density.
Description: Change from Baseline at Day 29 of the dosing period (start of AeroVanc/Placebo administration is considered Day 1 of the dosing period) in the number of MRSA colony forming units (CFU) in sputum culture.
Time Frame: Day 29 of treatment period
Population: Modified ITT population, which included all randomized patients who received any amount of study drug and had at least one scheduled post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Log10 CFU/mL
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 17 | 17 | 15 | 22
Log10 CFU/mL | -0.25 (0.181) | -0.30 (0.182) | -0.63 (0.232) | 0.16 (0.201)

2. Secondary Outcome: Change From Baseline in MRSA Sputum Density.
Time Frame: Day 8 of treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log10 CFU/mL
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 20 | 17 | 24 | 22
Log10 CFU/mL | -0.27 (0.208) | -0.28 (0.223) | -1.04 (0.193) | 0.08 (0.200)

3. Secondary Outcome: Change From Baseline in MRSA Sputum Density.
Time Frame: Day 15 of treatment period
Population: Modified ITT (MITT) population, which included all randomized patients who received any amount of study drug and had at least one scheduled post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Log10 CFU/mL
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 19 | 16 | 19 | 22
Log10 CFU/mL | -0.55 (0.259) | 0.09 (0.279) | -1.14 (0.229) | 0.26 (0.216)

4. Secondary Outcome: Change From Baseline in FEV1
Description: Absolute change from baseline in FEV1 percent predicted
Time Frame: Day 29 of treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FEV1
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 18 | 17 | 16 | 21
percentage of predicted FEV1 | 0.53 (1.343) | 1.15 (1.356) | -0.68 (1.1449) | -2.61 (1.314)

5. Secondary Outcome: Change From Baseline in FVC
Description: Absolute change from baseline in FVC percent predicted
Time Frame: Day 29 of treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FVC
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 18 | 17 | 16 | 21
percentage of predicted FVC | -0.07 (1.273) | 1.67 (1.283) | -0.47 (1.594) | -2.48 (1.423)

6. Secondary Outcome: Change From Baseline in Cystic Fibrosis Respiratory Symptom Diary (CFRSD-CRISS) Scores
Description: Change from Baseline in Cystic Fibrosis Respiratory Symptom Diary (CFRSD) Chronic Respiratory Infection Symptom Scores (CRISS). The minimum score is 0 and the maximum is 100, where a higher score means a worse outcome.
Time Frame: Day 29 of treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 17 | 17 | 17 | 21
score on a scale | -6.59 (2.620) | -3.02 (2.614) | -0.55 (2.701) | -5.43 (2.552)

7. Secondary Outcome: Time From Start of Dosing to First Administration of Other Antimicrobial Medications (Oral, Intravenous and/or Inhaled) Due to Respiratory Symptoms.
Time Frame: Entire study: Day 1 of treatment period through 8 week post-treatment follow up visit
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 20 | 20 | 24 | 23
days | 69.5 [34.0 to 107.0] | 80.0 [23.0 to NA] — 95% CI not calculable because 50% of patients were censored at time of study completion. | 48.0 [14.0 to 66.0] | NA [43.0 to NA] — Median and 95% CI not calculable because more than 50% of patients were censored at time of study completion.

8. Secondary Outcome: Time From Start of Dosing to Exacerbation of Signs/Symptoms (Fuchs Criteria).
Time Frame: Entire study: Day 1 of treatment period through 8 week post-treatment follow up visit
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 20 | 20 | 24 | 23
days | 107.0 [13.0 to 107.0] | NA [13.0 to NA] — Median and 95% CI not calculable because more than 50% of patients were censored at time of study completion. | 49.0 [14.0 to 84.0] | NA [37.0 to NA] — Median and 95% CI not calculable because more than 50% of patients were censored at time of study completion.

9. Secondary Outcome: Change From Baseline in High Sensitivity CRP
Time Frame: Day 29 of the dosing period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 17 | 17 | 15 | 22
mg/dL | -0.34 (0.132) | -0.18 (0.130) | 0.15 (0.223) | -0.09 (0.184)

10. Secondary Outcome: Change From Baseline in Blood Neutrophils
Time Frame: Day 29 of the dosing period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
Number analyzed (Participants) | 17 | 17 | 16 | 21
10^9 cells/L | 0.20 (0.569) | 1.23 (0.561) | -0.29 (0.557) | 0.04 (0.487)

ADVERSE EVENTS:
Arm/Group | AeroVanc 32 mg | Placebo to 32 mg | AeroVanc 64 mg | Placebo to 64 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/20 | 2/20 | 1/24 | 4/23
Other Adverse Events (participants affected / at risk) | 18/20 | 18/20 | 20/24 | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroVanc 32 mg (N=20) | Placebo to 32 mg (N=20) | AeroVanc 64 mg (N=24) | Placebo to 64 mg (N=23)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 (3) | 2 (3) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroVanc 32 mg (N=20) | Placebo to 32 mg (N=20) | AeroVanc 64 mg (N=24) | Placebo to 64 mg (N=23)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 7 (12) | 9 (11) | 10 (11)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (5) | 7 (7) | 7 (8)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 6 (6) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 5 (6) | 3 (3)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3) | 4 (4) | 1 (2)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Fatigue (General disorders) | 5 (6) | 4 (6) | 8 (8) | 3 (3)
Exercise tolerance decreased (General disorders) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 (3) | 5 (5) | 5 (5) | 2 (2)
Forced expiratory volume decreased (Investigations) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 4 (6) | 1 (1) | 2 (2) | 1 (1)
Sinus headache (Nervous system disorders) | 4 (4) | 1 (1) | 2 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Product taste abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peak expiratory flow rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No